CLINICAL TRIAL: NCT05889936
Title: A Transdiagnostic Intervention for Health-related Habits (LEV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Douglas Sjowall, Principal investigator, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The LEV Project
Record Dates: First submitted 2023-03-12; First posted 2023-06-05 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Intervention; Life Style; Health-Related Behavior; Feasibility; Quality of Life; Disabilities Physical; Disability Physical; Mental Health Wellness
MeSH Terms: conditions — Health Behavior | interventions — Levamisole

STUDY DESIGN:
Intervention Model Description: Feasibility trial with pre, peri and post measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with the Lev-intervention (Experimental): Screening of health-related habits using Lev-s + a three step/session intervention including the standard Lev protocol. Typically given over 10-20 weeks.
  Interventions: Behavioral: Lev

INTERVENTIONS:
Behavioral: Lev — Lev includes three sessions using psychoeducation, motivational interviewing, and applied behavioral analyses. Lev also include two homework assignments. The second session can be repeated if needed. Lev-s and Lev are described in two manuals.

SUMMARY:
Research problem and specific questions: Health-related habits influences mental and physical health. Still, screening and treatment of health-related habits, which can help to remedy health problems, is not done at all or very superficially. National guidelines emphasize the importance of prioritizing health-related habits, but there is a lack of implemented models. To solve this, the investigators have developed a transdiagnostic, interprofessional material intended for several care settings.

Study 1: Is LEV a feasible intervention in different healthcare contexts? Study 2: A functional roadmap to healthier habits: A thematic analysis of themes form the functional analysis of unhealthy and healthy lifestyle behavior in adults with disabilities This study will use data from study 1.

DETAILED DESCRIPTION:
Lev is a brief, transdiagnostic, interprofessional intervention targeting health-related habits that is intended for several care settings.This study will therefore be open for participants recruited from several types of healthcare services in Sweden.

Study 1: The feasibility trial investigates the following questions:

1. Eligibility to participate - how many of the healthcare workers that had received training in Lev started using it within 6 months? How many participants that were offered Lev agreed to take part in the intervention?
2. What were the reasons for not taking part or not completing Lev? Healthcare workers administering Lev will ask the declining participants for reasons to not take part in the intervention.
3. How many sessions and homework assignments did the participants complete? Lev includes screening (Lev-s), three sessions and two pre-specified home assignments. The administrating healthcare worker fills in completed sessions and assignments in the case report form. We will set the time limit to 6 months to complete the three sessions including all homework assignments.
4. Were there any differences between healthcare professions regarding how the applied behavioral analysis was performed (e.g., were there any differences regarding strategies suggested to the participant)?

   During session 2, a functional behavioral analysis is performed to generate strategies to help the participant reach their goal. The investigators will conduct a thematic analysis to identify themes for each healthcare profession administrating Lev. This will answer questions regarding if it is possible to conduct this type of analysis in Lev or if further adjustments are needed.
5. Level of acceptability: Was Lev perceived as creditable and satisfactory by healthcare workers and participants? Treatment credibility will be measured before Lev and after the last session for both participants and healthcare workers. Treatment satisfaction will be evaluated after each session and after the intervention is completed. Session evaluations will be done by both participants and healthcare workers.
6. Was there any part of Lev that was perceived less satisfactory by participants and healthcare workers? A thematic analysis (Braun et al., 2004) will be performed to extract what was perceived as useful and to identify areas of improvement. This will be done both for participants and the healthcare workers.
7. Do the intervention lead to adverse events?
8. Do Lev lead to healthier habits?
9. To what extent were individual goals met?
10. Did Lev lead to increased quality of life?

Study 2:

1. What general themes underlying unhealthy and healthy habits can be found in individuals with disabilities?
2. How do themes vary for specific living habits?
3. How do themes vary for specific disabilities?
4. How do themes for questions b and c vary depending on sex?

ELIGIBILITY:
Inclusion Criteria:

* Study 1 and 2 will include both adults with and without disabilities recruited from different healthcare contexts.

Exclusion Criteria:

* Intellectual disability of the degree where the participant is not able to follow the protocol in Lev.
* Insufficient command of the Swedish language/ unable to understand the content.
* Severe psychiatric comorbidity that makes participation difficult (e.g. severe depression, severe suicidality, severe anxiety, ongoing psychosis, manic episode), other circumstances that could make participation hard (e.g. homelessness).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Study 1: Completion rate healthcare workers | 6 month after completing the training.
  how many of the healthcare workers that had received training in Lev started using it within 6 months
Study 1: Completion rate participants | 6 month after starting the screening
  How many of the participants that started using Lev (i.e., completing screening with Lev-s) completed Lev (i.e., completing, 2 out of 3 steps)
Study 1: Level of treatment credibility healthcare workers | Immediately after the intervention (mean time 20 weeks)
  Was Lev perceived as creditable and by healthcare workers using Treatment and Credibility Scale. Four items for credibility and one for expectation on a 10 point Likert scale where higher values indicate higher credibility.
Study 1: Level of treatment credibility participants | Immediately after the intervention (mean time 20 weeks)
  Was Lev perceived as creditable and by participants using Treatment and Credibility Scale . Four items for credibility and one for expectation on a 10 point Likert scale where higher values indicate higher credibility.
Study 1: Treatment satisfaction healthcare workers (individual sessions) | Immediately after completing session 1. An average of 1-2 months from baseline
  Treatment satisfaction will be evaluated after session 1 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. The content of this session feels relevant
  2. The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist
  3. Is there something else you would like to add?
Study 1: Treatment satisfaction healthcare workers (individual sessions) | Immediately after completing session 2. An average of 2-4 months from baseline
  Treatment satisfaction will be evaluated after session 2 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. The content of this session feels relevant
  2. The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist
  3. Is there something else you would like to add?
Study 1: Treatment satisfaction healthcare workers (individual sessions) | Immediately after completing session 3. An average of 4-8 months from baseline
  Treatment satisfaction will be evaluated after session 3 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. The content of this session feels relevant
  2. The degree of difficulty in conveying the content of the session is at a reasonable level for me as a therapist
  3. Is there something else you would like to add?
Study 1: Treatment satisfaction participants (individual sessions) | After completing the first module in Lev. An average of 1-2 months from baseline
  Treatment satisfaction will be evaluated after session 1 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. After the meeting today, my knowledge of how I can change my lifestyle have increased.
  2. I will benefit from what we talked about during the meeting today
  3. The content of the meeting felt relevant based on my own experiences
  4. I understood the advice and strategies I was given that will help my change mine lifestyle habits
  5. I feel confident in how to use the advice and strategies
  6. I will use the advice and strategies
  7. I was listened to, the therapist understood my situation
  8. I was involved and helped to come up with suggestions for how I can reach my goals
  9. Is there something else you would like to add?
Study 1: Treatment satisfaction participants (individual sessions) | After completing the second module in Lev. An average of 2-4 month from baseline
  Treatment satisfaction will be evaluated after session 2 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. After the meeting today, my knowledge of how I can change my lifestyle have increased.
  2. I will benefit from what we talked about during the meeting today
  3. The content of the meeting felt relevant based on my own experiences
  4. I understood the advice and strategies I was given that will help my change mine lifestyle habits
  5. I feel confident in how to use the advice and strategies
  6. I will use the advice and strategies
  7. I was listened to, the therapist understood my situation
  8. I was involved and helped to come up with suggestions for how I can reach my goals
  9. Is there something else you would like to add?
Study 1: Treatment satisfaction participants (individual sessions) | After completing the third module in Lev. An average of 4-8 month from baseline
  Treatment satisfaction will be evaluated after session 3 using a modified version of the Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. After the meeting today, my knowledge of how I can change my lifestyle have increased.
  2. I will benefit from what we talked about during the meeting today
  3. The content of the meeting felt relevant based on my own experiences
  4. I understood the advice and strategies I was given that will help my change mine lifestyle habits
  5. I feel confident in how to use the advice and strategies
  6. I will use the advice and strategies
  7. I was listened to, the therapist understood my situation
  8. I was involved and helped to come up with suggestions for how I can reach my goals
  9. Is there something else you would like to add?
Study 1: Treatment satisfaction participants (the whole intervention) | Directly after completing the last treatment module in LEV (approximately at 10 weeks)
  Treatment satisfaction will be evaluated after competing the whole intervention using Patient Evaluation Questionnaire including 5 levels where higher levels indicate higher satisfaction.
  1. As a whole, the Lev has been clearly focused on how I can live healthier
  2. My knowledge of how I can have healthier habits has increased
  3. I can better deal with problems connected to my health-related habits
  4. I have had the opportunity to contribute opinions during the Lev
  5. I would consider participating in a similar interventions in the future
  The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Study 1: Open answer questions regarding Treatment satisfaction measured by The Evaluation Questionnaire | Directly after completing the last treatment module in LEV (approximately at 20 weeks).
  The treatment satisfaction questionnaire also included open questions that will be analyses using a qualitative thematic approach including the following questions:
  1. I feel that participating in Lev helped me in these ways
  2. How could the Lev have been better?
  3. What could I have done differently myself?
  4. Is there anything else you would like to add?
  A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.
Study 1: Well-being before and after the intervention measures by The Evaluation Questionnaire | Directly after completing the last treatment module in LEV (approximately at 20 weeks)
  ("How would you rate your well-being prior to the intervention?", "How would you rate your current well-being") at T1 and T2 on a scale 1-10 (1= very poor, 10= very good)
Study 1: Adverse events after the intervention | During the intervention up to week approximately week 20.
  Adverse events will be defined as spontaneous oral complaints or instances when patients stated that they experienced negative or unwanted effects during the intervention period.
  Serious adverse events will be defined as events that involved hospital care/hospitalization, etc. due to the intervention.
Study 2: What general themes underlying unhealthy and healthy habits can be found in individuals with disabilities? | During the second step in Lev (Approximately at 5-10 weeks)"
  Healthcare workers are instructed to enter what strategies they gave to the participant. Strategies from step 2 (page 16 workbook). The themes are extracted based on answers to the following two questions:
  This is what others can do to help me: ....... I can do this myself:...
  A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.

SECONDARY OUTCOMES:
Study 1: Quality of life measured with WHOQOL-BREF. | Before and after taking part in Lev (after is approximately at 10-20 weeks
  Is Quality of life affected when completing Lev? The intervention group fill in WHOQOL-BREF at baseline and follow-up. 5 level scale where high levels indicate higher quality of life.
Study 1: Do Lev lead to healthier habits? | Before and after taking part in Lev (after is approximately at 10-20 weeks
  The Lev-s will be used to measures living habits before and after taking part in Lev. The scale includes 4 levels where higher levels indicate healthier habits.
Study 1: To what extent were individual goals met? | After completing the whole intervention (approximately at 10-20 weeks
  During session 1 in the intervention, individual goals are set. The healthcare worker assesses to what extent the goals have been met using the goal attainment scale. 5 point scale where high vales indicate that goals have been reached to a higher extent.
Study 2: How do the themes (e.g., situation, context, behavior, short term gratification) behind unhealthy habits vary for specific living habits? | During the second step in Lev (Approximately at 5-10 weeks)
  To understand what what underlying behavior and situations that underlies specific unhealthy habits investigators will conduct exploratory qualitative thematic analysis.
  A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.
Study 2: How do the themes behind unhealthy habits vary for different disabilities? | During the second step in Lev (Approximately at 5-10 weeks)
  To understand what underlying behavior and situations that underlies unhealthy habits in different groups of disabilities we will conduct exploratory qualitative thematic analysis.
  A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.
Study 2: How do the themes behind unhealthy habits vary depending on sex? | During the second step in Lev (Approximately at 5-10 weeks)
  To understand if underlying behavior and situations that underlies unhealthy habits differ depending on sex we will conduct the thematic analysis also separately for sexes.
  A qualitative, thematic analysis will be performed to identify more general themes. There is not a template or scale to extract the themes. One rater suggest categories based on the similarity of answers. Another rater organizes the answers in the suggested themes. To be considered a theme, there must be over 85% similarity between raters.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sjöwall, PhD, Principal Investigator — Regions Stockholm; Joakim Lavesson, Bachelor, Study Chair — Region Stockholm
Locations (1):
- Region Stockholm, Habilitering & Hälsa, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Douglas Sjöwall will be responsible for granting access to data only to researchers who are participating in the publications for study 1 and 2.

REFERENCES:
- [Derived] Sjowall D, Brar A, Fladvad A, Langh U, Hirvikoski T. Feasibility trial of a transdiagnostic individual lifestyle evaluation and intervention (Lev-i) for health behavior change. PLoS One. 2026 Jan 12;21(1):e0339500. doi: 10.1371/journal.pone.0339500. eCollection 2026. PMID 41525256